CLINICAL TRIAL: NCT06711445
Title: Reliability of Tele-assessment of the Performance Tests in Patients With Knee Osteoarthritis
Brief Title: Tele-assessment of the Performance Tests in Patients With Knee Osteoarthritis
Acronym: Teleassessment
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Gülşah ÖZSOY, Assistant Professor, Selcuk University
Other Study IDs: SELCUKU_PT_GO_001
Record Dates: First submitted 2024-11-22; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Telerehabilitation; Tele-assessment; Knee Arthritis Osteoarthritis; Performance Measures
Keywords: Knee osteoarthritis; reliability; single leg stance test; tele-assessment; thirty second chair stand test; timed up and go test
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tele- assessment Group: The participants were evaluated in two settings on different days (24-48 h apart): (i) in clinical settings (face-to-face) and (ii) at home via 'WhatsApp' phone application (both asynchronized and synchronized tele-assessment).
  Interventions: Other: Tele-assessment

INTERVENTIONS:
Other: Tele-assessment — The participants were evaluated in two settings on different days (24-48 h apart): (i) in clinical settings (face-to-face) and (ii) at home via 'WhatsApp' phone application (both asynchronized and synchronized tele-assessment).
  The evaluations steps were as follows:
  1. Face-to-face/ Clinic assessment: Rater 1 completed all clinical assessments.
  2. Synchronized tele-assessment: Rater 1 repeated the same evaluations via video calls to the patients (these were recorded to be used in step 3).
  3. Asynchronized tele-assessment: Rater 2 evaluated the recordings of the remote evaluations (made in step 2).
  4. Retest of synchronized tele-assessment: Rater 1 evaluated patients via video calls (these were recorded to be used in step 5).
  5. Retest of asynchronized tele-assessment: Rater 2 evaluated the recordings of the remote evaluations (made in step 4).

SUMMARY:
The COVID-19 pandemic widely affected delivery mode of healthcare services. While fewer number of patients were allowed to attend face-to-face rehabilitation sessions, some services were totally unavailable due to the safety measures. The COVID-19 crisis highlighted the value and accelerated the improvement of "tele-assessment and tele-rehabilitation" applications. Consequently, reliable remote assessment approaches were required to evaluate the effectiveness of the remote programs. While tests such as TUG, SLS, and 30CST are valid and reliable for clinical use in patients with knee OA, their psychometric properties are yet to be investigated when used as tele-assessment tests. Therefore, this study aimed to examine the intra- and inter-rater reliability of the TUG, SLS, and 30CST as remote tests in patients with knee OA.

DETAILED DESCRIPTION:
As the main cause of disability and loss of function in lower limb in middle-aged to elderly individuals , knee osteoarthritis (OA) is the most common OA worldwide and its prevalence increases with age and obesity . Among non-pharmacological methods, which are the first line of knee OA treatment , physical therapy is commonly prescribed to alleviate pain and improve physical function. However, not all patients with knee OA have access to face-to-face rehabilitation sessions under direct supervision of physicians or physiotherapists. Thanks to telemedicine, patients' access to real-time communication with health professionals has been considerably facilitated in recent years.

Detailed and comprehensive assessment is a fundamental factor for an effective rehabilitation program. Different assessment tools are available to assess the effectiveness of rehabilitation in patients with knee OA. To assess physical performance, practical tests, which are time- and space-effective, such as Timed Up and Go Test (TUG), Thirty Second Chair Stand Test (30CST), and Single Leg Stance Test (SLS) are commonly used in patients with knee OA .COVID-19 crisis highlighted the value and accelerated the improvement of "tele-assessment and tele-rehabilitation" applications. Consequently, reliable remote assessment approaches were required to evaluate the effectiveness of the remote programs.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2 and 3 knee OA on the Kellgren and Lawrence (K/L) scale,
* radiologically confirmed
* pain in the knee,
* willingness to join the study

Exclusion Criteria:

* Grade 0, 1 and 4 knee OA on the K/L scale,
* central or peripheral nervous system involvement,
* previous knee surgery within the past six months,
* neurological or musculoskeletal disorders that would limit their performance on the tests,
* history of systemic arthritic conditions

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We used convenience sampling method to recruit patients diagnosed with knee OA by their medical doctor according to the guidelines of American College of Rheumatology (ACR).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Timed up and go test (TUG) | 2 days
  The TUG is a simple practical test that measures the time an individual needs to stand up from a standard chair, walk 3 meters at normal speed, turn around, walk back to the chair, and sit down. Our participants performed 3 trials and their best score (in seconds) was recorded as the primary outcome. Participants had at least 4 minutes of seated rest intervals between the trials. Before and after each test, fatigue and dyspnea (using Borg scale), and hemodynamic (heart rate and SpO2) were evaluated.
Single Leg Stance Test (SLS) | 2 days
  The participants used their leg with arthritic knee (in cases of unilateral involvement) or the more symptomatic leg (in cases of bilateral involvement) as the stance limb. The test was terminated when the free leg/foot touched the ground, or if excessive trunk/upper body movements (e.g., swinging arms) were observed. Participants were allowed to repeat the test if they scored less than10 seconds during the first attempt. If needed, participants could rest between the trials for recovery. Before and after each test, fatigue and dyspnea (using Borg scale), and hemodynamics (heart rate and SpO2) were evaluated.
Thirty second chair stand test (30 CST) | 2 days
  The 30 CST checks the number of repetitions in 30 seconds that an individual can stand up from a standard chair (not using the arms/hands, feet flat on the ground) and sit back again. Our test chair was 43 cm in height and had no armrest. The participants performed 3 trials and their best score was recorded as the test result. If needed, they were allowed to rest (>5 min) between the trials for recovery. Before and after each test, fatigue and dyspnea (using Borg scale), and hemodynamics (heart rate and SpO2) were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Gulsah Ozsoy, PhD, Study Chair — Selcuk University
Locations (1):
- Selcuk University, Faculty of Health Sciences, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takacs J, Carpenter MG, Garland SJ, Hunt MA. Test re-test reliability of centre of pressure measures during standing balance in individuals with knee osteoarthritis. Gait Posture. 2014;40(1):270-3. doi: 10.1016/j.gaitpost.2014.03.016. Epub 2014 Mar 27. PMID 24746407
- [Background] Gill S, Hely R, Page RS, Hely A, Harrison B, Landers S. Thirty second chair stand test: Test-retest reliability, agreement and minimum detectable change in people with early-stage knee osteoarthritis. Physiother Res Int. 2022 Jul;27(3):e1957. doi: 10.1002/pri.1957. Epub 2022 May 19. PMID 35592902
- [Background] Alghadir A, Anwer S, Brismee JM. The reliability and minimal detectable change of Timed Up and Go test in individuals with grade 1-3 knee osteoarthritis. BMC Musculoskelet Disord. 2015 Jul 30;16:174. doi: 10.1186/s12891-015-0637-8. PMID 26223312
- [Background] Hatfield GL, Morrison A, Wenman M, Hammond CA, Hunt MA. Clinical Tests of Standing Balance in the Knee Osteoarthritis Population: Systematic Review and Meta-analysis. Phys Ther. 2016 Mar;96(3):324-37. doi: 10.2522/ptj.20150025. Epub 2015 Jul 16. PMID 26183586
- [Background] French HP, Hager CK, Venience A, Fagan R, Meldrum D. Psychometric properties and domains of postural control tests for individuals with knee osteoarthritis: a systematic review. Int J Rehabil Res. 2020 Jun;43(2):102-115. doi: 10.1097/MRR.0000000000000403. PMID 32282571